CLINICAL TRIAL: NCT07063914
Title: Acceptability and Feasibility of a Stratified-Care School-Based Intervention for Adolescent Suicidal Ideation in Chile: A Study Protocol
Brief Title: Stratified-Care School-Based Intervention for Adolescent Suicidal Ideation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: University of Talca (Other); Fundación Crecer y Sanar (Unknown)
Responsible Party: Principal Investigator, Jorge Gaete, Full Professor, Universidad de los Andes, Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FCS2025
Record Dates: First submitted 2025-06-25; First posted 2025-07-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Suicidal Ideation
Keywords: suicide; adolescents; depression; schools; prevention
MeSH Terms: conditions — Suicidal Ideation; Suicide; Depression

STUDY DESIGN:
Intervention Model Description: This is an initial feasibility and a single-arm study with pre-post assessments and follow-ups at 3, 6, 9, and 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm with the stratified-care intervention Reframe-IT and CARIBOU (Other): single arm
  Interventions: Behavioral: Reframe-IT and CARIBOU

INTERVENTIONS:
Behavioral: Reframe-IT and CARIBOU — Reframe-IT+ An individual intervention based on cognitive-behavioral therapy (CBT) focused on developing skills in behavioral activation, cognitive restructuring, emotion regulation, stress tolerance, and problem-solving. It is delivered in the school setting by a trained psychologist from the research team. The program consists of 13 weekly sessions of 45 minutes each: 5 face-to-face sessions and 8 combined digital/in-person sessions where students use a computer under the supervision of a psychologist facilitator.
  CARIBOU An individual CBT-based intervention focused on behavioral activation, cognitive restructuring, problem-solving, and communication skills. It is conducted in the school setting by a trained psychologist and consists of 16 weekly sessions of 45 minutes each.

SUMMARY:
Background. Suicidal ideation and depressive symptoms are highly prevalent among adolescents, with suicide representing a leading cause of death in this age group worldwide. School-based indicated prevention programs using cognitive behavioral therapy (CBT) have shown promise in addressing these mental health challenges. The Reframe-IT+ (Chile) and CARIBOU (Canada) programs are CBT-based, individually delivered interventions targeting adolescents at risk of suicide. This study aims to evaluate a culturally adapted stratified-care model using these two interventions, matched to depressive symptom severity.

Methods. This is a quasi-experimental, single-arm study with pre-post assessments and follow-ups at 3, 6, 9, and 12 months. Six secondary schools with high socioeconomic vulnerability in Santiago, Chile, will participate. Students with suicidal ideation and mild/moderate depressive symptoms (PHQ-9 < 20) will be offered Reframe-IT+, while those with severe symptoms (PHQ-9 ≥ 20) will be offered CARIBOU. Primary outcomes include the acceptability of CARIBOU, feasibility of the stratified-care model, and implementation fidelity. Secondary outcomes include reductions in suicidal ideation, depression, anxiety, hopelessness, and improvements in functioning, quality of life, behavioral activation, emotional regulation, and problem-solving skills.

Discussion. This protocol addresses the need for scalable, culturally sensitive interventions for adolescent suicide prevention in school settings. By evaluating both the process and early outcomes of a stratified-care approach, this study will generate valuable evidence to inform future large-scale effectiveness trials and policy development in adolescent mental health.

DETAILED DESCRIPTION:
Suicide among adolescents and young people is a highly prevalent global issue, with suicidal ideation reaching rates of approximately 18% and suicide attempts around 6% (1). According to the Global Burden of Diseases, Injuries, and Risk Factors Study (GBD), suicide ranks as the fifth leading cause of death among individuals aged 10 to 24 (2), with a mortality rate of 6.0 per 100,000 in this age group (3). Suicide mortality increases with age: 1.2 per 100,000 among those aged 10-14; 6.7 among those aged 15-19; and 10.6 among those aged 20-24 (3). In Latin America, suicide mortality rates surpass global averages, reaching 9.8 per 100,000, and in Chile, the rate is 7.2 per 100,000 (3).

Numerous risk factors are associated with suicide, including genetic, biological, psychological, and social factors (4,5). Each case of suicide is caused by a unique, dynamic, and complex interaction of these elements (4,5). However, depression remains the most frequently reported common factor (4). A recent literature review found that between 50-65% of suicide cases met criteria for depression (4). Regarding its broader impact, depressive symptoms are even more prevalent than suicidal ideation, with global rates of 43.9%, including mild, moderate, and severe cases (6). Moreover, the number of depression cases among adolescents has grown exponentially, with a 21.6% increase in total cases and a 19% increase in incidence compared to the 1990s (7). In Chile, adolescent depression is estimated to affect 8.3% of the population, yet fewer than half receive mental health care (8).

Secondary schools are recognized as appropriate, accessible, and effective settings for suicide (9) and depression prevention programs (10) for adolescents. School-based interventions offer broad reach and enable large-scale prevention efforts (9,10). Evidence shows that such programs improve suicide awareness and coping skills to reduce suicidal thoughts and attempts (9,11,12). However, indicated interventions-those targeting at-risk individuals with clinical or psychosocial approaches such as cognitive-behavioral therapy (CBT)-remain less common in school settings (13), despite their established efficacy in other contexts (13), underscoring the need for further research on their implementation in schools.

Two CBT-based programs have demonstrated effectiveness and safety in reducing suicidal ideation and depressive symptoms. Both are indicated interventions, meaning they target individuals already at risk and are delivered individually.

The Reframe-IT program, developed in Australia, targets behavioral activation, cognitive restructuring, emotion regulation, stress tolerance, and problem-solving skills (14). It includes eight digital sessions designed for delivery by school well-being staff (14). A pilot randomized controlled trial in Australia showed greater reductions in suicidal ideation, depression, and hopelessness among the intervention group than controls, although differences were not statistically significant due to insufficient statistical power (14). In Chile, the research team collaborated with the University of Talca for over four years to culturally adapt Reframe-IT, developing Reframe-IT+ by adding five face-to-face sessions to the original eight. An initial pilot study with 52 participants showed high acceptability and reductions of 15.2 points in suicidal ideation and 3.5 in depressive symptoms (15). A subsequent RCT with 1,546 screened students and 100 randomized participants demonstrated significant decreases of 6.7 points in suicidal ideation and 3.1 in depressive symptoms (16). Following these positive results, a scaled-up quasi-experimental study in Santiago (CEC2024061) included 75 students and showed preliminary reductions of 2.5 points in suicidal ideation and 3.2 in depressive symptoms.

The CARIBOU program, developed in Canada, targets behavioral activation, cognitive restructuring, problem-solving, and communication skills (17). It consists of 16 sessions facilitated by trained professionals from diverse backgrounds. A non-randomized pilot study showed a 2-point reduction in depressive symptoms (17). Moreover, 80% of participants reported program engagement, and facilitators achieved 95% fidelity in implementation (17). The research team has initiated contact with Dr. Darren Courtney, CARIBOU's lead developer, to begin its cultural adaptation in Chile as part of the present study.

This study proposes a stratified-care intervention model in which treatment intensity is matched to individual needs, ensuring appropriate levels of care. Adolescents with suicidal ideation will be offered Reframe-IT+ if they present with mild or moderate depressive symptoms, and CARIBOU if they present with severe symptoms.

METHODOLOGY General Objective The general objective of this study is to examine the acceptability of the CARIBOU program and the feasibility and fidelity of implementing a stratified-care approach tailored to the needs of adolescents with suicidal ideation. Under this model, students with mild or moderate depressive symptoms (PHQ-9 < 20) will be offered the Reframe-IT+ program, and those with severe depressive symptoms (PHQ-9 ≥ 20) will be offered the CARIBOU program. Additionally, this study aims to explore the efficacy of a stratified-care intervention in adolescents at risk for suicide and with depressive symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for Educational Institutions

  * Located in Santiago, Chile.
  * Secondary education level (grades I-IV Medio).
  * Coeducational schools.
  * At least two classes per grade level in secondary education.
  * A minimum of 30 students per class.
  * Socioeconomic vulnerability level of ≥ 50%, as measured by the School Vulnerability Index (Índice de Vulnerabilidad Escolar - IVE-SINAE), which includes factors such as parental education and total household income.

Inclusion Criteria for Students

* Enrolled in grades I, II, or III Medio.
* Suicidal ideation within the past month, defined as a score ≥ 3 on the Columbia-Suicide Severity Rating Scale (C-SSRS).
* For the Reframe-IT+ program: mild or moderate depressive symptoms, defined as a PHQ-9 score < 20.
* For the CARIBOU program: severe depressive symptoms, defined as a PHQ-9 score ≥ 20.

Exclusion Criteria:

* Exclusion Criteria for Students

  * Participation in a structured suicide prevention program (Reframe-IT+) during 2024.
  * Severe psychotic symptoms, such as perceptual disturbances or delusional ideas, assessed during the eligibility interview.
  * Suicide attempt(s) in the past three months, assessed during the eligibility interview.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the CARIBOU Program | immediately post-intervention
  Acceptability will be assessed by examining how well the intervention is received by student participants and facilitators, and how well it addresses the needs of the target population. Upon completion of the program, participants will complete a general acceptability questionnaire and a module-specific acceptability questionnaire. Facilitators will complete a general acceptability questionnaire as well. All instruments were developed by the research team and are designed to measure the program's content in detail.
  Additionally, the Client Satisfaction Questionnaire (CSQ-8) will be used to assess overall satisfaction with the intervention (19). The CSQ-8 consists of 8 Likert-scale items with four response options, and includes open fields for comments and suggestions. It has demonstrated high internal consistency (α = 0.83-0.93) (20) and will be slightly adapted to reflect the context of this study.
Feasibility Recruitment | through study completion, an average of 1 year
  We will record the recruitment and characteristics of the sample
Feasibility Attendance to eligibility interviews | through study completion, an average of 1 year
  We will record the number of adolescents and families who attend eligibility interviews.
Feasibility Response rates to questionnaires | through study completion, an average of 1 year
  Response rates to questionnaires.
Feasibility Session attendance | through study completion, an average of 1 year
  Session attendance and progress through the program.
Feasibility Attrition | through study completion, an average of 1 year
  Participant retention and dropout rates.
Implementation Fidelity | through study completion, an average of 1 year
  Fidelity will be assessed by determining facilitator adherence to program protocols (Reframe-IT+ and CARIBOU). After each session, facilitators will complete a self-report monitoring form to record implementation fidelity. These forms were developed by the research team and assess the delivery of each session's content.

SECONDARY OUTCOMES:
Suicidal ideation | pre-post assessments and follow-ups at 3, 6, 9, and 12 months.
  Columbia Suicide Severity Rating Scale (C-SSRS): A six-item self-report instrument designed to assess the severity of suicidal ideation (21). The first 5 items explore the presence of suicidal ideation, intent, and planning during the past month. The sixth item explores suicidal behavior either as preparation, initiation of a suicide attempt, or a suicide attempt itself during the past three months. Each item is scored 0= "No" or 1= "Yes". The total score can range from 0 to 6 points. According to the answers given to the different items, categories of severity of suicidal ideation are established: If you answer "Yes" to item 1 and/or item 2, and "No" to all other items, a slight risk is indicated. If one answers "Yes" to item 3 and 'No' to all other items, a moderate risk is indicated, and finally, if one answers "Yes" to any of items 4, 5 and 6, a severe risk is indicated (21). It has high levels of internal consistency (α=0.73) (21). We will use a Spanish version previously validat
Suicidal ideation frecuency | pre-post assessments and follow-ups at 3, 6, 9, and 12 months.
  Suicidal Ideation Questionnaire-Junior (SIQ-JR). It is a 15-item self-report instrument designed to assess the frequency of suicidal ideation in children and adolescents during the past month (23). Each item is scored by Likert scale from 0="Never" to 6="Almost every day". The total score can range from 0 to 90 points. It is considered that a score > 30 points could imply a potential risk of suicide (23). It has high levels of internal consistency (α=0.91) and test-retest reliability (K=0.89) (23). We will use a Spanish version previously validated in adolescents in Chile, which showed high levels of reliability (ω =0.97) (24).
Depressive symptoms | pre-post assessments and follow-ups at 3, 6, 9, and 12 months.
  The Patient Health Questionnaire (PHQ-9). It is a nine-item self-report instrument designed to assess the frequency of depressive symptomatology (25). Each item is scored by Likert scale from 0="Never" to 3="Almost every day". The total score can range from 0 to 27 points. The interpretation is made by adding the total of the 9 questions as follows: 0-4 points, no depression; 5-9, mild depression; 10-14, moderate depression; 15-19, moderately severe depression; 20-27, severe depression (25). It has high levels of internal consistency (α=0.89) (25). We will use a Spanish version previously validated in adolescents in Chile, which showed high levels of reliability (α =0.78) (26).
Anxiety symptoms | pre-post assessments and follow-ups at 3, 6, 9, and 12 months.
  The Generalized Anxiety Disorder Questionnaire (GAD-7). It is a seven-item self-report instrument designed to assess the frequency of anxious symptomatology (27). Each item is scored by Likert scale from 0="Never" to 3="Almost every day". The total score can range from 0 to 21 points. The interpretation is made by adding the total of the 9 questions as follows: 0-4 points, no anxiety; 5-9, mild anxiety; 10-14, moderate anxiety; 15-21, severe anxiety (27). It has high levels of internal consistency (α=0.92) (27). We will use a Spanish version previously validated in adolescents in Chile, which showed high levels of reliability (α =0.86) (28).
Hopelessness | pre-post assessments and follow-ups at 3, 6, 9, and 12 months.
  Beck Hopelessness Scale (BHS): It is a 20-item self-report instrument designed to assess hopelessness (29). Each item is scored from 0="False" to 1="True". The total score can range from 0 to 20 points. Interpretation is done by summing the total of the 20 questions as follows: 0-3 points, asymptomatic; 4-8, mild hopelessness; 9-14, moderate hopelessness; 15-20, severe hopelessness. It has high levels of internal consistency (α=0.93) (29). We will use a Spanish version previously validated in young people in Chile, which showed high levels of reliability (α =0.86) (30).
Mood | pre-post assessments and follow-ups at 3, 6, 9, and 12 months.
  Mood and Feelings Questionnaire (Short version)(33). It is a self-report instrument designed to assess mood. It consists of 13 items that are answered on a Likert scale of 0= "Not true" and 2= "True". The total score can range from 0 to 26 points. Different studies have shown that it is a unidimensional scale in populations aged 6 to 18 years in girls and boys (34, 35). It has high levels of internal reliability (α = 0.80 to 0.91) and validity in cohorts of children aged 8-16 (33).
Psychotic symptomatology | pre-post assessments and follow-ups at 3, 6, 9, and 12 months.
  Community Assessment of Psychotic Experiences Scale (CAPE-P15) (31). It is a self-report instrument designed to assess psychotic symptomatology. It consists of 15 items that are answered on a Likert scale from 1 = "Never" to 4 = "Very often". Scores can range from 15 to 60 points. The scale assesses three domains: paranoid ideation (PI, 5 items), bizarre experiences (EB, 7 items), and perceptual abnormalities (PA, 3 items) (35). The questionnaire can be evaluated through critical item review, where for example perceptual disturbances with psychotic features can be considered with scores ≥ 3 on item 13, 14 or 15. In a validation study of a Chilean population of adolescents between 13 and 18 years of age, the trifactorial nature of the scale was confirmed. The internal reliability for these factors was 0.78 for IP; 0.84 for EB; and 0.88 for AP (32).
Impairment | pre-post assessments and follow-ups at 3, 6, 9, and 12 months
  Columbia Functional Impairment Scale (Youth Version)(36). It is a 13-item self-report instrument designed to assess the level of impairment in functioning in children and adolescents. Each item is scored on a scale from 0 = "No problem" to 4 = "Very big problem." The total score can range from 0 to 52 points. It has high levels of internal consistency, and the original study reported values of α = 0.70 to 0.78 across multiple assessment items (36). We have authorization from the authors of the scale to use the Spanish version.
Behavioral Activation | pre-post assessments and follow-ups at 3, 6, 9, and 12 months
  Behavioral Activation Scale for Depression (BADS) (37). It is a self-report instrument that explores different coping mechanisms in adolescents and adults. It has 25 items distributed in 4 subscales: Behavioral Activation, Avoidance/Rumination, Impaired Work/School functioning, and Impaired Social functioning. Each item is scored on a scale from 0 = "Strongly Disagree" to 6 = "Strongly Agree". The total score can range from 0 to 150 points. It has good levels of internal consistency, both for the total scale (α= 0.79), and for the subscales: Behavioral Activation (α = 0.87), Avoidance/Rumination (α = 0.83), Work/Ecological Impairment (α = 0.78) and Social Impairment (α = 0.83). It has been used in other Latin American countries (38), and we will use the Chilean version, which has been validated and shows good internal reliability indices (Behavioral Activation, α = 0.81; Avoidance/Rumination, α = 0.85; Work/Ecological Impairment, α = 0.81; and Social Impairment, α = 0.87)(39).
Problem-solving | pre-post assessments and follow-ups at 3, 6, 9, and 12 months
  Brief Problem Solving Inventory (SPSI-R). This 25-item self-report instrument was designed to assess problem solving in children and adolescents (40). It has two adaptive dimensions of problem solving (positive problem orientation and rational problem solving) and three dysfunctional dimensions (negative problem orientation, impulsivity/neglect style, and avoidance style). Each item is scored by Likert scale from 0="Not at all true for me" to 4="Extremely true for me". The total score can range from 0 to 100 points. It has high levels of internal consistency in all its scales (α=0.76 to 0.92) (40). It has been previously used in young people in Chile, which showed high levels of reliability (α =0.90) (41).
Emotion regulation | pre-post assessments and follow-ups at 3, 6, 9, and 12 months
  Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA). This 10-item self-report instrument was designed to assess problem solving in children and adolescents (42). It has an adaptive dimension of emotional regulation (cognitive reappraisal, 6 items) and a dysfunctional dimension (emotional suppression, 4 items). Each item is scored by Likert scale from 1="Strongly disagree" to 5="Strongly agree". The score for the cognitive reappraisal scale can range from 6 to 30 points and the score for the emotional suppression scale can range from 4 to 20 points. It has high levels of internal consistency the cognitive reappraisal (α=0.75) and emotional suppression subscales 0.82) (42). We will use a Spanish version previously validated in adolescents in Chile, which showed acceptable levels of reliability in the cognitive reappraisal (ω=0.76; α=0.76) and emotional suppression (ω=0.71; α=0.71) subscales (43).
Wellbeing and quality of life | pre-post assessments and follow-ups at 3, 6, 9, and 12 months
  KIDSCREEN-10 Index, Child and Adolescent Version (Kidscreen-10 Index). This 10-item self-report instrument was designed to assess well-being and health-related quality of life (44). It is a brief version of the Kidscreen-52 and the Kidscreen-27 (44). Each item is scored by Likert scale from 1="Never" to 5="Always". The total score can range from 10 to 50 points (44).It has high levels of internal consistency (α=0.82) (44). We will use a brief Spanish version previously validated in adolescents in Chile, which showed high levels of reliability (α =0.89) (45).

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Gaete, MD. PhD., Study Director — Universidad de Los Andes
Locations (1):
- Universidad de los Andes, Santiago, Las Condes, Chile

IPD SHARING:
Plan to Share IPD: No
the data will have personal information of minors

REFERENCES:
- [Background] Lim KS, Wong CH, McIntyre RS, Wang J, Zhang Z, Tran BX, Tan W, Ho CS, Ho RC. Global Lifetime and 12-Month Prevalence of Suicidal Behavior, Deliberate Self-Harm and Non-Suicidal Self-Injury in Children and Adolescents between 1989 and 2018: A Meta-Analysis. Int J Environ Res Public Health. 2019 Nov 19;16(22):4581. doi: 10.3390/ijerph16224581. PMID 31752375